CLINICAL TRIAL: NCT00160056
Title: The Effect of Antecedent Hypoglycaemia on β2-adrenergic Sensitivity in Subjects With Homozygous Arg16 and gly16 Polymorphism of the β2-adrenergic Receptor
Brief Title: The Effect of Antecedent Hypoglycaemia on β2-adrenergic Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: HB2-001
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes; Hypoglycemia Unawareness
Keywords: Hypoglycemia unawareness; Diabetes; adrenal receptor; adrenerg respons; adrenergic beta-agonists; salbutamol
MeSH Terms: conditions — Diabetes Mellitus | interventions — Hig1 protein, mouse

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Hypoglycemia (Other): Intrerfvention is a hypoglycemic stimulus
  Interventions: Procedure: Hypoglycemia

INTERVENTIONS:
Procedure: Hypoglycemia

SUMMARY:
Hypoglycaemia unawareness is a common complication in patients with type 1 diabetes and with insulin-treated type 2 diabetes of long duration. The loss of autonomic symptoms to hypoglycemia does not solely depend on loss of adrenaline responses.Differences in sensitivity to catecholamines may also be involved.

Reconciling the data on β2-adrenergic receptor polymorphism to those on loss of β-adrenergic sensitivity in diabetic patients with hypoglycemia unawareness, we hypothesize that hypoglycemia unawareness is at least partly the result of desensitization of the β2-adrenergic receptor and that patients who are homozygous for arginine at codon 16 are particularly susceptible for this desensitization process, whereas patients who are homozygous for glycine at codon 16 are resistant for desensitization.

Objectives

1. To determine whether, and if so to what extent, antecedent hypoglycemia reduces β2-adrenergic sensitivity in healthy subjects with Arg16 homozygosity.
2. To investigate whether or not healthy subjects with Gly16 homozygosity are resistant to desensitization
3. To confirm that antecedent hypoglycemia reduces the heart rate response to isoproterenol and to assess to what extent this reduced response is mediated by impairments in baroreflex sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Homozygous for Arginine at codon 16 or homozygous Gly at codon 16
* No regular usage of medication other than oral contraceptives

Exclusion Criteria:

* History of cerebrovascular, cardiovascular, or peripheral vascular disease
* Smoking
* Alcohol usage of more than 10 units per week
* Inability to abstain from xanthine-derivatives (coffee, tea, cola, chocolate, cacao) or alcohol for 2 days
* BMI above 30 kg/m2
* Participation to any other trial in the preceding 3 months
* Ongoing disease of any kind
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Smits, PhD, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Schouwenberg BJ, Smits P, Tack CJ, de Galan BE. The effect of antecedent hypoglycaemia on beta(2)-adrenergic sensitivity in healthy participants with the Arg16Gly polymorphism of the beta(2)-adrenergic receptor. Diabetologia. 2011 May;54(5):1212-8. doi: 10.1007/s00125-011-2062-3. Epub 2011 Feb 6. PMID 21298412